CLINICAL TRIAL: NCT01255332
Title: Efficacy of Helicobacter Pylori Eradication for the 1st Line Treatment of Immune Thrombocytopenic Purpura (ITP) Patients With Moderate Thrombocytopenia
Brief Title: Helicobacter Pylori Immune Thrombocytopenic Purpura
Acronym: HpyloriITP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: COSAH, Cooperative Study Group A for Hematology
Other Study IDs: C-023
Record Dates: First submitted 2010-11-24; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-11

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- C13-urea breath test: positive: lansoprazole 30mg bid, amoxicillin 1000mg bid and clarithromycin 500mg bid for 7 days

SUMMARY:
We designed a study for evaluate the efficacy of Helicobacter pylori eradication for the 1st line treatment of immune thrombocytopenic purpura (ITP) patients with moderate thrombocytopenia.

If this eradication treatment is revealed effective on ITP patients with more than 30X109/L of platelet, it would be valuable treatment especially for young ITP patients with mild to moderate thrombocytopenia.

DETAILED DESCRIPTION:
lansoprazole 30mg bid, amoxicillin 1000mg bid and clarithromycin 500mg bid for 7 days. (Jeil Pharm. CO. LTD. will provide lansoprazole.) C13-UBT, at 4 weeks after onset of treatment, to determine eradication

ELIGIBILITY:
Inclusion Criteria:

* 20~55 years old
* Persistent or chronic ITP patients, defined by international working group ( persistent: between 3 to 12 months from diagnosis, chronic: lasting for more than 12 months)
* 30X109/L ≤ platelet count ≤ 70X109/L
* C13-urea breath test: positive
* no previous ITP treatment
* no previous H. pylori eradication treatment
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* Patients who have any cause of thrombocytopenia such as HIV, HCV infection, lymphoproliferative disease, liver disease, definite SLE, drug, MDS, leukemia
* Uncontrolled hypothyroidism or hyperthyroidism
* Acute active bleeding or infection
* Who taking anti-coagulant or aspirin
* Patients with penicillin allergy
* Patients with side effects of macrolide.
* Patients who taking Mizolastine, Terfenadine, Cisapride, Pimozide, Astemizole, Ergot alkaloid and its derivatives (Ergotamine, Dihydroergotamine), Bepridil, or Atazanavir
* Patients who have known allergy or severe side effect on study drugs
* Pregnant or lactating women
* Clinically relevant hepatic or renal disease (Creatinine clearance ≤ 30mL/min)
* patients who cannot understand informed consent or express his/her condition

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: immune thrombocytopenic purpura
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Overall response | 2 years
  Overall response rate at 3 months after treatment

SECONDARY OUTCOMES:
Eradication rate of H. pylori | 2 years
  We designed a study for evaluate the efficacy of Helicobacter pylori eradication for the 1st line treatment of immune thrombocytopenic purpura (ITP) patients with moderate thrombocytopenia.
  * Duration of response
  * Side effect and safety of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hee Lee, professor, Principal Investigator — Asan Medical Center; Hyo Jung Kim, professor, Principal Investigator — Department of Internal Medicine, Hallym University Sacred Heart Hospital
Locations (1):
- Asan Medical Center, Seoul, Asanbyeongwon-gil, Songpa-gu, South Korea

REFERENCES:
- [Derived] Kim H, Lee WS, Lee KH, Bae SH, Kim MK, Joo YD, Zang DY, Jo JC, Lee SM, Lee JH, Lee JH, Kim DY, Ryoo HM, Hyun MS, Kim HJ; CoOperative Study Group A for Hematology (COSAH). Efficacy of Helicobacter pylori eradication for the 1st line treatment of immune thrombocytopenia patients with moderate thrombocytopenia. Ann Hematol. 2015 May;94(5):739-46. doi: 10.1007/s00277-014-2268-9. Epub 2014 Dec 13. PMID 25501820
- See also: Efficacy of Helicobacter pylori eradication, anti-D and danazol combination in steroid dependant or refractory immune thrombocytopenia (ITP) — http://www.google.co.kr